CLINICAL TRIAL: NCT05501782
Title: Evaluation of Intuitive Eating and Hedonic Hunger Status and the Effects of Intuitive Eating and Hedonic Deficit on Body Mass Index, Mental Health and Sleep Quality in University Students.
Brief Title: Evaluation of Intuitive Eating and Hedonic Hunger in University Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gülin Öztürk Özkan, Head of department (PhD) Assistant Professor, Istanbul Medeniyet University
Other Study IDs: 2022/0145
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: INTUITIVE EATING; Hedonic Hunger
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — A questionnaire consisting of seven parts was applied to the participants. In the first part, 20; demographic data and general health status of the participants; There were 11 questions including nutritional habits and anthropometric measurements (body weight and height). The other parts of the questionnaire were the Intuitive Eating Scale (IES-2), Power of Food Scale (PFS-Tr), Food Craving Questionnaire (FCQ-T), the Pittsburg Sleep Quality Scale (PUKI), Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) and Palatable Eating Motive Scale (PEMS), respectively contains. Consent from the participants was also obtained with the questionnaire form.

SUMMARY:
This study was conducted with the participation of 62 female and 38 male students between the ages of 18-36 studying at various universities. A questionnaire consisting of seven parts was applied to the participants. In the first part, 20; demographic data and general health status of the participants; There were 11 questions including nutritional habits and anthropometric measurements (body weight and height). The other parts of the questionnaire were the Intuitive Eating Scale (IES-2), Power of Food Scale (PFS-Tr), Food Craving Questionnaire (FCQ-T), the Pittsburg Sleep Quality Scale (PUKI), Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) and Palatable Eating Motive Scale (PEMS), respectively contains. Consent from the participants was also obtained with the questionnaire form.

ELIGIBILITY:
Inclusion Criteria:

* University students who agreed to participate in the study

Exclusion Criteria:

* University students who did not want to participate in the study baby and kids elderly adolescents pregnant women breastfeeding mothers

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students who agreed to participate in the study
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Intuitive eating scale (IES-2) | 2 months
  Intuitive eating scale (IES-2) consists of 23 questions, each of which includes five options ranging from strongly agree to strongly disagree. A 5-point Likert scale was used in the scale. In 1,2,3,7,8,9,10 questions, strongly disagree 5, disagree 4, undecided 3, agree 2 and strongly agree 1 point. The scoring of the answers to the other questions is in the opposite order (strongly disagree 1, disagree 2, undecided 3, agree 4, and strongly agree 5 points). The scale score was calculated by dividing the total score obtained at the end of the questions by 23. Intuitive eating behavior also increases in parallel with the increase in the scale score. The median values of the Intuitive Eating Scores of the students participating in the study were found. Participants with a scale score below the median value were considered as having no intuitive eating behavior, and participants with a median value and above were considered individuals with intuitive eating behavior
Power of food scale (PFS) | 2 months
  Power of food scale (PFS) is a scale developed to evaluate the effects of palatable foods on the psychological and hedonic states of individuals. The Turkish version with a reliability study was used in this study (PFS-Tr) A validated version of this scale consisting of 15 items was used. The scale was evaluated using a 5-point Likert scale. Accordingly, I strongly disagree 1 point, I disagree 2 points, I am undecided 3 points, I agree 4 points, and I strongly agree 5 points. The scores obtained from all items were divided into five and the scale score was found. It was concluded that the hedonic hunger levels of individuals with a nutritional power score of 2.5 and above increased. It has been accepted that individuals with a high score are sensitive to the food environment and psychologically under the influence of food
Food Craving Questionnaire (FCQ) | 2 months
  Food Craving Questionnaire (FCQ) is a scale developed for the assessment of food cravings. The Turkish version with a reliability study was used in this study (FCQ-T). In this scale, evaluation is made with a 6-point Likert scale. It was scored always 6 points, mostly 5 points, often 4 points, occasionally 3 points, rarely 2 points, never 1 point. High scale scores of the participants indicate an increase in food cravings
Pittsburg Sleep Quality Scale (PUKI) | 2 months
  Pittsburg Sleep Quality Scale (PUKI) is a scale developed to evaluate sleep quality. This scale includes 18 items with 7 components. These components are subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime sleep dysfunction. Each component is scored between 0-3 points, with a maximum total score of 21. A total score of 5 or more indicates poor sleep quality, and an increase in the score indicates a decrease in sleep quality
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) | 2 months
  the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS), whose reliability study was conducted, was used. The scale consists of 14 questions and is evaluated with a 5-point Likert scale. It is scored as 1 point to strongly disagree, 2 points to disagree, 3 points to slightly agree, 4 points to agree and 5 points to completely agree. The total score on the scale is between 14 and 70. The increase in the total score indicates that the mental well-being of the individual increases.